

# Brief Group Intervention Based on Acceptance and Commitment Therapy (ACT) for Problem Gambling: A Pilot Study

ID: 2025-81

Document Date: February 23, 2025

Principal Investigators: Francisco Montesinos, Ph.D. – David Lobato, Ph.D.

**Participant Information Sheet and Informed Consent** 

#### **Study Title**

Brief Group Intervention Based on Acceptance and Commitment Therapy (ACT) for Problematic Gambling: A Pilot Study

#### **Promoter**

Universidad Europea de Madrid

### **Principal Investigator**

Francisco Montesinos, Ph.D. - David Lobato, Ph.D.

# **Collaborating Investigator**

Rubén Pérez Pérez

#### **Faculty**

Faculty of Biomedical and Health Sciences, Universidad Europea de Madrid

#### Introduction

You are being invited to participate in a research study aimed at Spanish-speaking adults who engage in gambling activities (e.g., sports betting, poker, blackjack, slot machines, roulette) and wish to change this behavior and improve their psychological well-being.

This study has been approved by the Research Ethics Committee of the Hospital Universitario de Getafe and the Spanish Agency of Medicines and Medical Devices, in accordance with current legislation (Royal Decree 1090/2015 and European Regulation 536/2014).

Please read this information carefully. If you have any questions, you may contact:

Dr. Francisco Montesinos: francisco.montesinos@universidadeuropea.es

Dr. David Lobato: david.lobato@universidadeuropea.es

Mr. Rubén Pérez: ruben.perez@universidadeuropea.es

# **Voluntary Participation**

Your participation is entirely voluntary. You may choose not to participate or withdraw at any time without any consequences or impact on future services.

# **Study Objective**

To evaluate the feasibility and acceptability of a brief online group psychological program based on psychological flexibility, aimed at helping individuals dissatisfied with their gambling behavior to manage it more effectively and improve their psychological wellbeing.

# **Study Description**

The study includes:

1. Initial Assessment: An interview and questionnaires to determine eligibility.

- 2. Intervention: An 8-session online group therapy based on ACT, led by a licensed psychologist.
- 3. Follow-up: Completion of questionnaires at baseline, post-intervention, and at 3 and 6 months follow-up.

#### **Study Activities Timeline**

Total Duration: Approximately 33 weeks

Weeks 1–9: Initial assessment and 8 weekly group sessions (90 minutes each)

Weeks 21 & 33: Follow-up assessments

#### **Risks and Discomforts**

There are no anticipated risks. The intervention is evidence-based and has shown benefits in reducing gambling behavior and improving emotional well-being. All activities are conducted online.

# **Participant Responsibilities**

- Complete all questionnaires honestly and privately
- Submit weekly data on gambling behavior and emotional state
- Attend all sessions in a private setting
- Maintain confidentiality and respect for other participants
- Notify the therapist of any emotional difficulties or absences
- Avoid starting other psychological treatments without prior consultation

#### **Potential Benefits**

- Development of skills to manage gambling behavior
- Improved emotional well-being
- Contribution to scientific research and future treatment development

#### **Pregnancy Warning**

Participation poses no risk in the event of pregnancy.

#### **Alternative Treatments**

If you choose not to participate, you may seek help from public addiction services or associations such as APEAP or AJER.

#### Insurance

The study promoter has an insurance policy in accordance with Royal Decree 1090/2015 to cover any harm related to participation.

#### **Data Protection**

Your data will be anonymized and handled in compliance with Spanish data protection laws (LOPD 3/2018). Only authorized personnel will access your data, and it will not be used to identify you.

# **Costs and Compensation**

Participation is free of charge and conducted online, so no travel or additional expenses are required.

# **Additional Information**

The study is registered at https://www.clinicaltrials.gov/. Any relevant new information will be shared with you during the study.

| Informed Consent Form I, |
|---|
| $\square$ Have read the information sheet |
| $\square$ Have had the opportunity to ask questions |
| $\square$ Have received sufficient information |
| □Have spoken with |
| $\square$ Understand that participation is voluntary |
| $\square$ Understand I can withdraw at any time without explanation or impact on my care |
| I freely consent to participate in this study. |
| Participant Signature |
| Date: / / |